CLINICAL TRIAL: NCT05876741
Title: Validation of Prognostic Accuracy of ABC ( Age, Blood Urea Nitrogen , Co-morbidities ) and Horibe Pre-endoscopy Scoring Systems in Patients With Upper Gastrointestinal Bleeding in Sohag University Hospital .
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Aly, Resident of Tropical medicine and gastroenterology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-04-09MS
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Upper GI Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Vital Signs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: patient presented with hematemesis , coffee ground vomiting , melena and haematoectasia to gastroenterology department will be included.
  Interventions: Diagnostic Test: history taking , vital signs and labaratory investigations

INTERVENTIONS:
Diagnostic Test: history taking , vital signs and labaratory investigations — 1. Complete history taking:
     With stress on age, sex, epigastric pain, comorbidities (ischemic heart disease, diabetes, liver cirrhosis, renal failure, malignancy), syncope, disturbed conscious level, blood transfusion, drug history .
  2. Clinical examination:
     Pulse, blood pressure, calculating the shock index, pallor, jaundice, cachexia, purpura, ecchymosis, conscious level, abdominal examination.
  3. Laboratory investigations:
     * Complete blood count (CBC).
     * Creatinine and blood urea nitrogen (BUN).
     * liver function tests (serum bilirubin, serum albumin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), prothrombin time (PT), prothrombin concentration (PC), and international normalized ratio (INR)).
     * Serum electrolytes and arterial blood gases.
     * Fasting blood sugar.
  4. Assessment of risk and predicting outcomes by:
     * Pre-endoscopic Rockall score (pRS).
     * Glasgow-Blatchford score (GBS).
     * AIMS65 score.
     * ABC score.
     * Horibe score.

SUMMARY:
Upper gastrointestinal bleeding (UGIB) is a common medical emergency with significant morbidity and mortality. Treating physicians are urged to perform rapid diagnosis, careful risk assessment, and effective resuscitation to improve outcomes and limit the risk of complications .

Several prognostic scoring systems have been developed to identify high- and low-risk patients presenting with UGIB and are commonly used in emergency departments to classify patients. Identifying low-risk patients who can be treated electively or on an outpatient basis can reduce the burden on physicians, patients, and the healthcare system (Rout et al., 2019). On the other hand, identifying high-risk patients who require immediate hospitalization and intervention can help avoid delays in treatment, thereby reducing morbidity and mortality. By using appropriate risk assessment tools, it is possible not only to predict which patients are at risk of adverse events such as rebleeding or death, but also to make management decisions such as the timing of endoscopy, length of hospital stay, and level of care .

Several pre-endoscopy scoring systems have been developed to predict the need for hospital-based intervention (transfusion, endoscopic treatment, radiological embolization, or surgery) and 30-day mortality risk. The pre-endoscopic Rockall score (pRS), the Glasgow-Blatchford score (GBS), and the AIMS65 score are the most widely used scoring systems in clinical practice .

The GBS was established as a tool for assessing the need for medical interventions (e.g., blood transfusion, therapeutic endoscopy, or surgery). The pRS and AIMS65 have been shown to predict mortality most accurately among patients with UGIB. In addition, AIMS65 is a simple risk score consisting of easily accessible parameters that was created to improve adherence to risk stratification and facilitate early triage and targeted therapy. However, there are limitations in these scoring systems. The GBS is difficult to calculate in routine clinical practice due to its complex nature . Moreover, the discriminative performance of existing scores for the prediction of mortality is relatively poor .

Two new relatively simple scores were developed to predict the outcome in patients presenting with UGIB, the Horibe gastrointestinal bleeding (HARBINGER) score (Horibe et al., 2016), and the Age, Blood tests, and Comorbidities (ABC) score (Laursen et al., 2021). The Horibe score was developed primarily to triage patients presented with UGIB (need for hospital admission, endoscopic intervention), while the ABC score was developed to predict 30-day mortality in patients presenting with UGIB. Both scores demonstrated good performance in studies conducted for their validation and may be superior to the existing pre-endoscopy scores .

ELIGIBILITY:
Inclusion Criteria:

* All patients presented to the outpatient clinic, emergency or inpatient section of the Tropical Medicine and Gastroenterology Department, Sohag University Hospital by UGIB as defined by haematemesis (vomiting of blood or coffee ground emesis), or melena will be included in the study.

Exclusion Criteria:

* · Patients less than 18 years.

  * Missed follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presented to the outpatient clinic, emergency or inpatient section of the Tropical Medicine and Gastroenterology Department, Sohag University Hospital by UGIB as defined by haematemesis (vomiting of blood or coffee ground emesis), or melena will be included in the study.
  Exclusion Criteria:
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
comparison between old and new upper git bleeding scoring systems regarding accuracy and prognostic value . | 1 monthe
  As UGIB is a medical emergency requiring timely decisions, physicians must know exactly which risk scores are reliable for each clinical outcome. The currently existing scores are either difficult to calculate or not accurate at predicting the outcome for which they developed. Two new scores (the Horibe and the ABC) were developed to overcome the drawbacks of the existing scores, So, we conducted the current study to validate them.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horibe M, Iwasaki E, Bazerbachi F, Kaneko T, Matsuzaki J, Minami K, Masaoka T, Hosoe N, Ogura Y, Namiki S, Hosoda Y, Ogata H, Chan AT, Kanai T. Horibe GI bleeding prediction score: a simple score for triage decision-making in patients with suspected upper GI bleeding. Gastrointest Endosc. 2020 Sep;92(3):578-588.e4. doi: 10.1016/j.gie.2020.03.3846. Epub 2020 Mar 30. PMID 32240682
- [Background] Horibe M, Kaneko T, Yokogawa N, Yokota T, Okawa O, Nakatani Y, Ogura Y, Matsuzaki J, Iwasaki E, Hosoe N, Masaoka T, Inadomi JM, Suzuki H, Kanai T, Namiki S. A simple scoring system to assess the need for an endoscopic intervention in suspected upper gastrointestinal bleeding: A prospective cohort study. Dig Liver Dis. 2016 Oct;48(10):1180-6. doi: 10.1016/j.dld.2016.07.009. Epub 2016 Jul 18. PMID 27507771
- [Background] Kim MS, Choi J, Shin WC. AIMS65 scoring system is comparable to Glasgow-Blatchford score or Rockall score for prediction of clinical outcomes for non-variceal upper gastrointestinal bleeding. BMC Gastroenterol. 2019 Jul 26;19(1):136. doi: 10.1186/s12876-019-1051-8. PMID 31349816
- [Background] Laursen SB, Oakland K, Laine L, Bieber V, Marmo R, Redondo-Cerezo E, Dalton HR, Ngu J, Schultz M, Soncini M, Gralnek I, Jairath V, Murray IA, Stanley AJ. ABC score: a new risk score that accurately predicts mortality in acute upper and lower gastrointestinal bleeding: an international multicentre study. Gut. 2021 Apr;70(4):707-716. doi: 10.1136/gutjnl-2019-320002. Epub 2020 Jul 28. PMID 32723845